CLINICAL TRIAL: NCT07055425
Title: The Role of Qmax/eGFR Ratio in Assessing Symptom Severity and QoL in Men Over 40 With LUTS
Brief Title: Association Between Qmax/eGFR Ratio and LUTS Severity in Men Over 40
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tarik Emre Sener, Assoc. Prof., Marmara University
Other Study IDs: MAR.UAD.0024
Record Dates: First submitted 2025-06-21; First posted 2025-07-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Lower Urinary Tract Symptom; Voiding Dysfunction; Male Urological Health; Renal Function; Benign Prostate Obstruction (BPO)
Keywords: Lower Urinary Tract Symptom; Benign Prostate Obstruction (BPO); Male Urological Health; Voiding Dysfunction; Aging Male
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men Over 40 With LUTS: Male patients aged 40 years or older presenting with lower urinary tract symptoms (LUTS), who undergo uroflowmetry and renal function testing, and complete the IPSS questionnaire. No interventions will be applied. This group will be prospectively observed for the association between Qmax/eGFR ratio and symptom severity.

SUMMARY:
This study will look at how well a measure called the Qmax/eGFR ratio is related to the severity of urination problems in men over the age of 40. Qmax is a test that shows how fast a person can urinate, and eGFR is a number that reflects kidney function. Men who have urinary symptoms will be asked to do a urine flow test, a blood test, and fill out a questionnaire about their symptoms and quality of life. We will study if there is a link between the Qmax/eGFR ratio and how severe their symptoms are. The results may help doctors better understand how kidney and urinary function are related in men with these problems.

DETAILED DESCRIPTION:
This prospective observational study aims to explore the clinical relevance of the Qmax/eGFR ratio in men over 40 years of age presenting with lower urinary tract symptoms (LUTS). Qmax, derived from uroflowmetry, reflects bladder emptying function, while eGFR represents renal filtration capacity. While both parameters are routinely measured in clinical practice, their combined predictive or associative value in LUTS severity has not been well defined.

Participants will undergo standard non-invasive assessments including uroflowmetry, serum creatinine testing (for eGFR calculation), and will complete the International Prostate Symptom Score (IPSS) questionnaire. The IPSS includes both total symptom score and quality of life (QoL) component. The primary objective is to evaluate the correlation between the Qmax/eGFR ratio and IPSS total score. Secondary objectives include the relationship between Qmax/eGFR and QoL scores, as well as analysis based on prostate volume categories.

This study seeks to identify whether the Qmax/eGFR ratio may serve as a composite marker reflecting both voiding efficiency and renal function in the clinical assessment of LUTS, potentially supporting more individualized decision-making in urological practice.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 40 years or older presenting with lower urinary tract symptoms (LUTS)
* Able to provide informed consent
* Willing and able to undergo uroflowmetry and blood testing
* Able to complete the IPSS questionnaire, including the QoL item
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m²

Exclusion Criteria:

* History of urological surgery (e.g., prostatectomy, bladder surgery)
* Diagnosed or suspected prostate cancer
* Active urinary tract infection (based on clinical symptoms or urinalysis)
* Neurological conditions affecting bladder function (e.g., Parkinson's disease, spinal cord injury)
* Presence of an indwelling urinary catheter at enrollment
* eGFR < 30 mL/min/1.73m²
* Inability to perform uroflowmetry or complete clinical evaluations

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male outpatients aged 40 years or older who present with lower urinary tract symptoms (LUTS) to the urology clinic. Participants will be evaluated during routine clinical visits and must be capable of completing symptom questionnaires and undergoing non-invasive tests such as uroflowmetry and blood sampling. The study population is drawn from a single tertiary academic medical center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Qmax/eGFR Ratio and Total IPSS Score | At baseline
  This outcome assesses the statistical correlation between the Qmax/eGFR ratio and the total International Prostate Symptom Score (IPSS). Pearson or Spearman correlation analysis will be used to evaluate the relationship between the ratio and LUTS severity.
Correlation Between Qmax/eGFR Ratio and IPSS Quality of Life Subscore | At baseline
  This outcome evaluates the correlation between the Qmax/eGFR ratio and the IPSS Quality of Life (QoL) subscore, aiming to assess the association between voiding/renal parameters and patient-perceived well-being.

SECONDARY OUTCOMES:
Factors Associated With Qmax/eGFR Ratio | At baseline
  This outcome aims to identify clinical factors that may influence the Qmax/eGFR ratio in men over 40 with lower urinary tract symptoms. Variables to be analyzed may include age, prostate volume, voided volume, and average flow rate (Qave), among others. Multivariable analysis will be performed to explore independent associations.
Association of Clinical Variables With Qmax/eGFR Ratio | At baseline
  This analysis will identify clinical parameters independently associated with Qmax/eGFR ratio, including age, prostate volume, voided volume, and average flow rate (Qave). Multivariable regression models will be used to determine significant predictors.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared due to the observational design, single-center setting, and the absence of genomic or identifying information. However, anonymized data may be made available upon reasonable scientific request and after appropriate ethical and institutional approvals.